CLINICAL TRIAL: NCT03577470
Title: Italian Retrospective and Prospective Observation of Antiretroviral Treatment in Patients Taking DarunavIr/cobicistAt Plus eMtricitabine and Tenofovir AlafeNamide fumaraTE - DIAMANTE
Brief Title: An Italian Observation of Antiretroviral Treatment in Participants Taking Darunavir/ Cobicistat Plus Emtricitabine and Tenofovir Alafenamide Fumarate
Acronym: DIAMANTE
Status: Completed | Type: Observational
Sponsor: Janssen-Cilag S.p.A. (Industry)
Responsible Party: Sponsor
Other Study IDs: CR108466; TMC114FD1HTX4011 (Other: Janssen-Cilag S.p.A., Italy)
Record Dates: First submitted 2018-06-07; First posted 2018-07-05 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Human Immunodeficiency Virus (HIV)
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — symtuza

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Group 1: Participants will not receive any intervention as a part of this study. This group will include participants in treatment with Darunavir/ Cobicistat/ Emtricitabine/ Tenofovir Alafenamide (D/C/F/TAF), who were always being treated with boosted-darunavir (DRV)-based regimen. The primary data source will be the medical records of each participant participating in this study.
  Interventions: Drug: D/C/F/TAF Fixed-Dose Combination (FDC)
- Group 2: Participants will not receive any intervention as a part of this study. This group will include participants who started their antiretroviral (ARV) treatment with any combination excluding DRV before starting D/C/F/TAF treatments, who were always being treated with ARV treatment with any combination excluding DRV before starting D/C/F/TAF treatments. The primary data source will be the medical records of each participant participating in this study.
  Interventions: Drug: D/C/F/TAF Fixed-Dose Combination (FDC)
- Group 3: Participants will not receive any intervention as a part of this study. This group will include participants started with D/C/F/TAF as naive. The primary data source will be the medical records of each participant participating in this study.
  Interventions: Drug: D/C/F/TAF Fixed-Dose Combination (FDC)

INTERVENTIONS:
Drug: D/C/F/TAF Fixed-Dose Combination (FDC) — Participants in treatment with D/C/F/TAF FDC, coming from different treatment histories will be observed in this study. No interventions will be administered as a part of this study.
  Other Names: Symtuza

SUMMARY:
The purpose of this study is to describe the effectiveness of Darunavir/ Cobicistat/ Emtricitabine/ Tenofovir Alafenamide (D/C/F/TAF), measured as virological response at Week 48 as per Food and Drug Administration (FDA) snapshot algorithm through collection of daily practice data in the Italian setting.

ELIGIBILITY:
Inclusion Criteria:

* Having a confirmed diagnosis of Human Immunodeficiency Virus-1 (HIV-1)
* Must sign a participation agreement/Informed Consent Form (ICF) allowing data collection and source data verification in accordance with local requirements
* Taking Darunavir/ Cobicistat/ Emtricitabine/ Tenofovir Alafenamide (D/C/F/TAF) as per Summary of Product Characteristics (SmPCs) since at least one month before enrollment:

  i) Experienced participants [Group 1 and 2]: a) started their antiretroviral (ARV) treatment not before 1/1/2015, b) having at least 1 year of ARV treatment history at study enrollment, c) Group 1, having always been treated with Darunavir (DRV) since the start of ARV treatment as naïve, d) Group 2, not having been treated with DRV before starting of D/C/F/TAF, ii.) Naive (any Viral Load (VL) participants (Group 3)

Exclusion Criteria:

* Participants unable to read, to write, to understand and sign the ICF
* Currently enrolled in an interventional study
* Currently enrolled in an observational study sponsored or supported by Janssen
* Chemotherapy scheduled during study observation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Any participant with confirmed diagnosis of Human immunodeficiency virus (HIV) infection will be enrolled and around 20 Infectious Diseases Centers in Italy will be involved.
Sampling Method: Non-Probability Sample
Enrollment: 246 (Actual)
Dates: Start 2018-06-13 (Actual); Primary Completion 2020-09-28 (Actual); Study Completion 2020-09-28 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants with Virological Response at Week 48 | At Week 48
  Percentage of participants with virologic response defined as plasma Human Immunodeficiency Virus-Ribonucleic Acid (HIV-RNA) Viral Load (VL) less than (<) 50 copies per milliliter (cp/mL) measured according to Food and Drug Administration (FDA) snapshot algorithm will be reported.

SECONDARY OUTCOMES:
Participant's Previous Antiretroviral (ARV) Treatment History Determined Using the Web-Based Electronic Case Report Form (eCRF) | At Baseline (Visit 1)
  Participants previous antiretroviral (ARV) treatment history will be determined using the web-based electronic case report form (eCRF) which will be prepared based on the study flow chart.
Time to Virosuppression | At Baseline (Visit 1)
  For participants entering with VL greater than (>) 50cp/mL, the time to virosuppression will be recorded.
Number of Participants with Detectability Below Level of Quantification <50 copies/mL | At Baseline (Visit 1)
  Number of participants with detectability below level of quantification <50 copies/mL will be reported.
Cluster Differentiation 4 (CD4) Cells Nadir Count | At Baseline (Visit 1)
  CD4 cells nadir count will be reported.
CD4 Cell Count | At Baseline (Visit 1)
  CD4 cells count will be reported.
Cluster Differentiation 4/ Cluster Differentiation 8 (CD4/CD8) Ratio | At Baseline (Visit 1)
  CD4/CD8 ratio will be reported.
Percentage of Participants with VL<50cp/mL Measured by the FDA Snapshot Algorithm and Stratified by Age | Up to Week 48
  The percentage of participants having virological response defined as plasma HIV-RNA VL< 50 cp/mL measured by the FDA snapshot algorithm, stratified by age [<50, greater than (>) 50 and < 65, > 65 years according to participants' number] will be reported.
Percentage of Participants with VL < 50 cp/mL Measured by the FDA Snapshot Algorithm and Stratified by Gender at Birth | Up to Week 48
  The percentage of participants having virological response defined as plasma HIV-RNA VL< 50 cp/mL measured by the FDA snapshot algorithm, stratified by gender at birth will be reported.
Percentage of Participants with VL < 50 cp/mL Measured by the FDA Snapshot Algorithm and Stratified by Original Group | Up to Week 48
  The percentage of participants having virological response defined as plasma HIV-RNA VL< 50 cp/mL measured by the FDA snapshot algorithm, stratified by original group will be reported.
Percentage of Participants Withdrawing From the Study for any Reason | Up to Week 48
  The percentage of participants withdrawing from the study for any reason will be reported.
Percentage of Participants who are Virologic Responders (VL<50 cp/mL) Measured by the Time to Loss of Virological Response (TLOVR) Algorithm | Up to Week 48
  The percentage of participants having virological response defined as VL< 50 cp/mL, measured by the TLOVR algorithm dataset will be reported. In the TLOVR dataset, participant responses at a specified threshold of HIV-1 RNA (<50 copies/mL) are determined by using the Food and Drug Administration's TLOVR algorithm. Using the TLOVR algorithm, participants are considered to have failed on therapy if they never achieved confirmed RNA levels below the threshold, if they had confirmed rebound of RNA above the threshold, if they made a non-permitted change in background regimen, or if they permanently discontinued investigational product for any reason.
Percentage of Participants with Virological Failure in Virosuppressed Participants | Up to Week 48
  Percentage of participants with virological failure (two consecutive measures of VL greater than or equal to (>=) 50cp/mL) in virosuppressed participants with virological rebound will be calculated and reported.
Change from Baseline in Human Immunodeficiency Virus-Treatment Satisfaction Questionnaire Score (HIV-TSQs) at Week 48 | Baseline and Week 48
  The HIV-TSQ is a 10-item self-reported scale that measures overall satisfaction with treatment by specific items that includes current treatment, control, side effects, demands, convenience, flexibility, understanding, lifestyle, recommend to others, continue. The HIV-TSQ items are summed up to produce a treatment satisfaction total score (0 to 60) and an individual satisfaction rating for each item (0 to 6). The higher the score, the greater the improvement in treatment satisfaction as compared to the past few weeks. A smaller score represents a decline in treatment satisfaction compared to the past few weeks. HIV-TSQs will be recorded onto paper forms and will be considered as source data.
Change from Baseline in Participants Reported Outcome Based on Narrative Plots at Week 48 | Baseline and Week 48
  Narrative plots will be recorded onto paper forms and will be considered as source data to describe the participants experience during treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen-Cilag S.p.A., Italy Clinical Trial, Study Director — Janssen-Cilag S.p.A.
Locations (18):
- Italy (18):
  - Azienda Ospedaliera Papa Giovanni XXIII, Bergamo
  - Azienda Ospedaliera Spedali Civili di Brescia, Brescia
  - ASST Valle Olona - P.O. di Busto Arsizio, Busto Arsizio
  - Ente Ospedaliero Ospedeli Galliera, Genova
  - Ospedale San Raffaele, Milan
  - Ospedale San Paolo Clinica Universitaria Malattie Infettive E Tropicali, Milan
  - A.O. Ospedale L. Sacco - Polo Universitario, Milan
  - Div Malattie Infettive - Ospedale L. Sacco, Milan
  - Azienda Ospedaliero Universitaria di Cagliari - Policlinico Duilio Casula di Monserrato, Monserrato
  - Azienda Ospedaliera dei Colli - P.O. 'D. Cotugno', Napoli
  - Azienda Ospedaliera di Padova, Padua
  - Azienda Ospedaliero Universitaria Policlinico Paolo Giaccone, Palermo
  - Policlinico Tor Vergata, Roma
  - Istituto nazionale malattie infettive 'L. Spallanzani', Roma
  - Universita Di Roma 'La Sapienza', Roma
  - Istituto di Ematologia - Clinica Universitaria, Sassari
  - A O Universitaria Senese Ospedale Santa Maria alle Scotte, Siena
  - Ospedale Amedeo di Savoia, Torino